CLINICAL TRIAL: NCT06344923
Title: Does Suturing the Peritoneum and Anterior Rectus Sheath Affect the Safety of Temporary Loop Ileostomy After Laparoscopic Anterior Rectal Resection
Brief Title: Peritoneum and Anterior Rectus Sheath Suturing and Ileostomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KYLL
Record Dates: First submitted 2024-03-24; First posted 2024-04-03 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-03

CONDITIONS: Ileostomy - Stoma; Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — Ileostomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified preventive ileostomy (Experimental): Ileostomy with a support rod instead of the layer of peritoneum and anterior rectus sheath suturing
  Interventions: Procedure: Ileostomy with a support rod instead of the layer of peritoneum and anterior rectus sheath suturing
- conventional preventive ileostomy (Active Comparator): Ileostomy with the layer of the peritoneum and anterior rectus sheath suturing
  Interventions: Procedure: Ileostomy with the layer of the peritoneum and anterior rectus sheath suturing

INTERVENTIONS:
Procedure: Ileostomy with a support rod instead of the layer of peritoneum and anterior rectus sheath suturing — The terminal ileum about 30cm proximal to the cecum was recognized and was lifted out of the body through the auxiliary incision at the right lower abdomen and made sure that the ileum was not twisted. Appropriate sutures can be used to narrow the peritoneal incision, preferably by inserting one finger. A support rod, made of a 24# silicone drainage tube with a 1ml syringe was passed through the mesentery of the small intestine. The support rod was removed two weeks after surgery. It is appropriate that the ileum wall protruded from the epidermis by about 3cm. After suturing trocar sites, the loop ileostomy was opened along the longitudinal axis of the intestinal wall, and 4-0 absorbable suture was used to fix the stoma and subcutaneous tissue circumferentially with 16-20 stitches.
  Arms: modified preventive ileostomy
Procedure: Ileostomy with the layer of the peritoneum and anterior rectus sheath suturing — The terminal ileum about 30cm proximal to the cecum was recognized and was lifted out of the body through the auxiliary incision at the right lower abdomen and made sure that the ileum was not twisted. Appropriate sutures can be used to narrow the peritoneal incision, preferably by inserting one finger. The seromuscular layer of the ileum or the mesentery was intermittently sutured with peritoneum and the anterior sheath of the rectus abdominis circumferentially with 8-10 stitches (3-0 silk thread). It is appropriate that the ileum wall protruded from the epidermis by about 3cm. After suturing trocar sites, the loop ileostomy was opened along the longitudinal axis of the intestinal wall, and 4-0 absorbable suture was used to fix the stoma and subcutaneous tissue circumferentially with 16-20 stitches
  Arms: conventional preventive ileostomy

SUMMARY:
In the era of laparoscopy, ileostomy via specimen extraction site has been proposed as a novel approach for temporary ostomy creation to prevent anastomotic leak after laparoscopic low anterior rectal resection. Whether suturing the layer of the peritoneum and anterior rectus sheath affects the safety of this novel approach has not been investigated.

ELIGIBILITY:
Inclusion Criteria:

* preventive ileostomy in laparoscopic rectal surgery

Exclusion Criteria:

* ileostomy due to anastomotic leak

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
postoperative complications related to ileostomy | after primary surgery to ileostomy closure (6 months after primary surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China